CLINICAL TRIAL: NCT03299270
Title: GOSAFE Study Geriatric Oncology Surgical Assessment and Functional rEcovery After Surgery An International Prospective Audit to Evaluate Postoperative Functional Outcomes and Quality of Life After Cancer Surgery in Geriatric Patients
Brief Title: Geriatric Oncology Surgical Assessment and Functional rEcovery After Surgery
Acronym: GOSAFE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AUSL ROMAGNA (Other)
Collaborators: European Society of Surgical Oncology (Other); International Society of Geriatric Oncology (Other); IRST (Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori) (Unknown)
Responsible Party: Sponsor-Investigator, AUSL ROMAGNA, Azienda USL della Romagna, AUSL Romagna Rimini
Organization: AUSL Romagna Rimini (Other)
Other Study IDs: GOSAFE
Record Dates: First submitted 2017-09-20; First posted 2017-10-03 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Elderly; Solid Malignancy
Keywords: Surgery; Solid malignancy; Elderly; Functional recovery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Elderly patiences with solid malignancy
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Quality of Life and Functional recovery questionnaires

SUMMARY:
Multicenter, international, prospective, observational study, designed to evaluate the postoperative results in terms of quality of life and functional recovery of elderly patients after major cancer surgery.

The global expected duration of the study is 3 years, during which cancer patients over 70 years old undergoing major surgery will be evaluated before and after the surgical intervention, at 30 days, 3- and 6-months follow-up. The study is non-for-profit. Given the observational nature of the study, the original treatment plan, as designed by each individual recruiting centre, will not be altered or affected by the study inclusion. Inclusion in the study does not imply any deviation from the current standard of practice, and no change is expected to the perioperative treatment at any point. Patients will be only asked to complete simple screening/assessment tests.

DETAILED DESCRIPTION:
GOSAFE study is a prospective international collaborative high-quality registry aiming to gain knowledge about postoperative outcomes in older cancer patients with a particular emphasis on QoL and FR. The target is to obtain meaningful data to assist clinicians in tailoring the care, avoiding under/over-treatment, providing robust data to identify new strategies to improve functional outcomes in older cancer patients.

Recruiting centers will collect data prospectively. Recruited patients will be followed for 6 months after their surgery.

The original treatment plan, as designed by each individual recruiting centre, will not be altered or affected by the study inclusion.

Centers should ensure that they would make every possible effort to include all consecutive eligible patients during the study period and provide completeness of data entry to ensure a 'real-life' study.

Patients both gender, both gender, aged ≥70, affected by solid malignancy undergoing elective major surgical procedures with curative or palliative intent are eligible.

Inclusion in the study does not imply any deviation from the current standard of practice, and no change is expected to the perioperative treatment at any point. Patients will be only asked to complete simple screening/assessment tests.

For every eligible patient, demographic data will be collected at baseline followed by a fast preoperative functional assessment. Data regarding surgical procedures and perioperative measures will be collected. Complications will be reported and graded according to Clavien-Dindo Classification. Three- and six-month follow up data will be collected after surgery within a range of 2 weeks from the due date.

The Full Analysis Set (FAS) consists of all registered patients. The primary endpoint will be measured for all registered subjects who fulfill preoperative and postoperative EQ VAS. Demographic and baseline patient characteristics will be summarized for all patients in the FAS. Continuous-scaled variables (e.g., age) will be summarized with means, medians, standard deviations, quartiles, and minimum and maximum values. Categorical variables (e.g., sex) will be summarized using patient counts and percentages. Study endpoints and variables will be evaluated using descriptive statistics, and the key figures of the distributions will be presented in tables. Univariate analyses will allow for a first overview of potentially influential factors.

Multiple linear regression models will be performed in order to evaluate predictors of functional recovery at 3 months and 6 months after surgery.

Exploratory subgroup analyses will be performed. Missing values will be replaced and estimated using multiple imputations. Furthermore, sensitivity analysis will be executed using complete-case analysis.

A sample size of 265 patients who completed pre and postoperative EQ VAS questionnaires will have a 90% power to detect an effect size of 0,2 between pre and post surgery ,using a paired t-test with a 0,05 two sided significance level.

Given a potential loss to follow-up (about 10%), uncompleted questionnaires (about 10%) and postoperative mortality (about 15%), the sample size will be increased to 350-400 patients (see ref 18 and 19).

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive patients, both gender, aged ≥70
2. Patients affected by solid malignancy
3. Patients undergoing elective major surgical procedures with curative or palliative intent (all major procedures including any resection, for any cancer, via any operative approach, open, laparoscopic, robotic, etc…)
4. Informed consent obtainment

Exclusion Criteria:

1. Patients undergoing emergent/urgent surgical procedures
2. Planned hospital stay less than 48 hours

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Centers should ensure that they would make every possible effort to include all consecutive eligible patients during the study period and provide completeness of data entry to ensure a 'real-life' study.
Sampling Method: Non-Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) | 6 months
  To evaluate the effects of surgery on patients' life perception by comparing pre- and post-operative QoL in elderly patients undergoing major surgery for solid malignancies using a self-reported Quality of Life assessment tool

SECONDARY OUTCOMES:
Functional recovery (FR) | 6 months
  To evaluate FR in terms of nutritional status, restoration of daily activities and cognitive status
Morbidity | 6 months
  To evaluate 3 and 6 months postoperative morbidity
Mortality | 6 months
  To evaluate 3 and 6 months postoperative mortality
Prognostic factors | 6 months
  To obtain prognostic factors for postoperative functional recovery which will assist in the treatment planning /intervention of future elderly patients who are offered surgery for cancer

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Giampaolo, MD, Principal Investigator — AUSL Romagna
Locations (28):
- United States (4):
  - Cleveland Clinic Florida, Weston, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Pennsylvenia Medical Center, Philadelphia, Pennsylvania
  - Roger William Medical Centre, Providence, Rhode Island
- Medical School, Aristotle University of Thessaloniki, Thessaloniki, Greece
- Rabin Medical Center, Petah Tikva, Israel
- Italy (13):
  - IstitutoTumori Giovanni Paolo II, Bari, Apulia
  - Ospedale di Forlì, Forlì, Forli-Cesena
  - Ospedale S. Andrea, Rome, Lazio
  - IRCCS Ospedale S. Martino Genova, Chirurgia Generale ad indirizzo oncologico, Genoa, Liguria
  - IRCCS Ospedale S. Martino Genova, Clinica Chirurgica 1, Genoa, Liguria
  - Humanitas, Rozzano, Milano
  - Ospedale di Desio, Desio, Monza E Brianza
  - Ospedale S. Matteo degli Infermi, Spoleto, Perugia
  - General Surgery Unit, Faenza, Ravenna
  - Ospedale di Riccione, Riccione, Rimini
  - Ospedale Niguarda, Milan
  - Ospedale di Piacenza, Piacenza
  - Clinica S. Rita, Vercelli
- Groeningen University Hospital, Groningen, Netherlands
- Institute of clinical medicine, Oslo, Norway
- Jagiellonian University Medical College, Krakow, Poland
- Portugal (2):
  - General Surgery dept,Hospital Sao Francisco Xavier (CHLO), Lisbon
  - Unidade Local de Saúde do Litoral Alentejano (ULSLA), Santiago do Cacém
- Spain (2):
  - Universidad Miguel Hernández. Elche. Alicante, Alicante
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (2):
  - Dept. of Surgical Oncology - St. Helens Hospital of Liverpool, Liverpool
  - Manchester Royal Infirmary, University of Manchester, Manchester